CLINICAL TRIAL: NCT01337011
Title: Pilot Study Comparing the Effect of Intra-coronary Versus Intramyocardial Application of Enriched CD133pos Autologous Bone Marrow Derived Stem Cells for Improving Left Ventricular Function in Chronic Ischemic Cardiomyopathy
Brief Title: Intra-coronary Versus Intramyocardial Application of Enriched CD133pos Autologous Bone Marrow Derived Stem Cells
Acronym: AlsterMACS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study was stopped due to funding issues
Sponsor: Asklepios proresearch (Industry)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1884; 2009-013103-63 (EudraCT Number)
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure
Keywords: Chronic Ischemic Cardiomyopathy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Comparison of the effect of CD133pos. bone marrow derived stem cells using the intra-myocardial vs. the intra-coronary route of administration for improving left ventricular function in patients with chronic ischemic cardiomopathy.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intra-coronary administration (Experimental): Application of stem cells using the intra-coronary route.
  Interventions: Other: autologous CD133pos stem cell application
- intra-myocardial administration (Experimental): Application of stem cells using the intra-myocardial route.
  Interventions: Other: autologous CD133pos stem cell application

INTERVENTIONS:
Other: autologous CD133pos stem cell application — The study aims to show efficacy of both intra-myocardial autologous CD133pos bone marrow cell application as well as intra-coronary CD133pos cell application in patients with symptomatic ischemic heart disease. In addition, efficacy between the two delivery routes will be compared.

SUMMARY:
This is a pilot study comparing the effect of intra-coronary versus intramyocardial application of enriched CD133pos autologous bone marrow derived stem cells for improving left ventricular function in chronic ischemic cardiomyopathy.

DETAILED DESCRIPTION:
Recent years have seen a tremendous improvement of possibilities to restore normal cardiac perfusion of the coronary arteries both by surgical and interventional techniques. In addition, several pharmacological approaches are available to block the mal-adaptive molecular signaling initiated by the Renin/Angiotensin/Aldosteron (RAAS) system. Device therapy achieving resychronisation has lowered morbidity and mortality. However, heart failure therapy still falls short to address the underlying disease of the heart muscle: loss of contractile force.

To achieve this aim and restore contractile force a regenerative approach is required. Early experimental studies suggested bone marrow cells to be able to differentiate towards functional cardiomyocytes when injected into the scar area after ischemic injury.2 These and other studies lead to clinical trials, where bone marrow cells were injected into the coronary circulation. Lately, the first completed multi-center, placebo-controlled, double-blinded study found several end points to be improved including global left ventricular function 3. At the same time genetically labelled experimental mouse models demonstrated differentiation of bone marrow cells towards a cardiomyocyte lineage to be a rare event,4 questioning at least the proposed molecular and cellular mechanism of intra-coronary cell therapy. Furthermore, several other clinical trials recently performed did either find no or a very limited effect of intra-coronary applied bone marrow cells. The effect appears to be related to improved angiogenesis. Our group has recently shown that in mammals endogenous regeneration of myocardium does occur after injury and can be enhanced via specific signaling pathways.5 Whether intra-coronary cell therapy is the ideal approach to enhance this process is currently unclear.

References:

1. Nieminen MS, Brutsaert D, Dickstein K, Drexler H, Follath F, Harjola VP, Hochadel M, Komajda M, Lassus J, Lopez-Sendon JL, Ponikowski P, Tavazzi L. EuroHeart Failure Survey II (EHFS II): a survey on hospitalized acute heart failure patients: description of population. Eur Heart J. 2006;27:2725-2736.
2. Orlic D, Kajstura J, Chimenti S, Limana F, Jakoniuk I, Quaini F, Nadal-Ginard B, Bodine DM, Leri A, Anversa P. Mobilized bone marrow cells repair the infarcted heart, improving function and survival. Proc Natl Acad Sci U S A. 2001;98:10344-10349.
3. Schachinger V, Erbs S, Elsasser A, Haberbosch W, Hambrecht R, Holschermann H, Yu J, Corti R, Mathey DG, Hamm CW, Suselbeck T, Assmus B, Tonn T, Dimmeler S, Zeiher AM, the R-AMII. Intracoronary Bone Marrow-Derived Progenitor Cells in Acute Myocardial Infarction. N Engl J Med. 2006;355:1210-1221.
4. Murry CE, Soonpaa MH, Reinecke H, Nakajima H, Nakajima HO, Rubart M, Pasumarthi KB, Virag JI, Bartelmez SH, Poppa V, Bradford G, Dowell JD, Williams DA, Field LJ. Haematopoietic stem cells do not transdifferentiate into cardiac myocytes in myocardial infarcts. Nature. 2004;428:664-668.
5. Zelarayan L, Noack C, Sekkali B, Kmecova J, Gehrke C, Renger A, Zafiriou MP, Nagel Rvd, Dietz R, Windt LJd, Balligand J-L, Bergmann MW. beta-catenin downregulation attenuates ischemic cardiac remodeling through enhanced resident precursor cell differentiation. Proc Natl Acad Sci U S A. 2008;105:19762-19767.
6. Krause KT, Jaquet K, Geidel S, Schneider C, Mandel C, Stoll HP, Hertting K, Harle T, Kuck KH. Percutaneous endocardial injection of erythropoietin: assessment of cardioprotection by electromechanical mapping. Eur J Heart Fail. 2006;8:443-450.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 80 years old
* Of female and male gender
* Patient has reduced ejection fraction as evaluated by routine clinical angiogram, echocardiography or MRI (≤45%) due to ischemic heart disease
* symptomatic heart failure NYHA ≥ II on optimal therapy
* coronary artery in the target region that can be used for cell infusion
* Patient has been informed of the nature of the clinical trial and agrees to its provision and has provided written informed consent

Exclusion Criteria:

* planned or performed CABG surgery or PCI within 4 weeks of study entry
* recent myocardial infarction (< 6 months)
* TIMI flow < II in the coronary artery selected for infusion
* cardiogenic shock requiring mechanical ventilation or intra-aortic balloon pump
* progressive tumor disease
* primary disease of bone marrow including mal-function of components of the coagulation system
* women of child-bearing age premenopausal
* LV wall thickness < 5mm at planned site of injection
* ventricular wall thrombus
* severe aortic valvular heart disease
* severe atrial or ventricular tachycardia unresponsive to intravenous or oral drug therapy
* aneurysm of the anterior wall
* history of stroke
* know diseases of the liver resulting in reduced plasmatic coagulation with spontaneous INR >2
* patients with chronic infectious diseases (HBV, HCV, HIV, seropositivity for Treponema pallidum)
* patients taking part or have taken part in other clinical trials within the past 3 months
* patients unable to provide informed consent
* any other medical condition that the enrolling physician deems significant in representing a potential hazard for the patient when participating in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2016-03-02 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
LVEF | after 6 to 12 months
  Improvement of global left ventricular function as well as global strain rate as assessed by echocardiography. Transthoracic echocardiography will be performed at baseline and after 6 and 12 month. Images are acquired in the standard parasternal and apical views.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bergmann, PD Dr., Principal Investigator — Asklepios Kliniken Hamburg GmbH
Locations (1):
- ASKLEPIOS Klinik St. Georg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No